CLINICAL TRIAL: NCT00859768
Title: The Effectiveness of the Screening Inventory of Psychosocial Problems (SIPP) in Cancer Patients Treated With Radiotherapy.
Brief Title: The Effectiveness of the Screening Inventory of Psychosocial Problems (SIPP) in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Netherlands Open University (Other)
Collaborators: Dutch Cancer Society (Other); Maastricht University Medical Center (Other); Institute Verbeeten (Other); Maastro Clinic, The Netherlands (Other)
Responsible Party: Lilian Lechner, PhD, Netherlands Open University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MB254; Dutch Cancer Society (Registry Identifier: 2008-4008)
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2009-03

CONDITIONS: Breast Cancer; Lung Cancer; Prostate Cancer; Bladder Cancer; Cervix Cancer; Cancer of Endometrium; Cancer of Skin; Non-Hodgkin Lymphoma; Colorectal Cancer
Keywords: Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Skin Neoplasms; Lymphoma, Non-Hodgkin; Colorectal Neoplasms; Neoplasms | interventions — Psychiatric Rehabilitation; Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention group 1 (Experimental): Pre-test measures are assessed. The patient receives the SIPP twice during their RT period. The first time is before the first consultation with the radiotherapist and the second time is before the last consultation at the end of the RT period. At both time points, the SIPP is handed over to the radiotherapist at the start of the consultation. The radiotherapist screens the scores of the SIPP to get an overview of potential psychosocial problems and patient's needs of psychosocial care. Follow-up measures are directly after first consultation (T2) and at three (T3) and twelve months (T4) after first measurement.
  Interventions: Other: Questionnaire administration
- Intervention group 2 (Experimental): No pre-test measures are assessed. The patient receives the SIPP twice during their RT period. The first time is before the first consultation with the radiotherapist and the second time is before the last consultation at the end of the RT period. At both time points, the SIPP is handed over to the radiotherapist at the start of the consultation. The radiotherapist screens the scores of the SIPP to get an overview of potential psychosocial problems and patient's needs of psychosocial care. Follow-up measures are directly after first consultation (T2) and at three (T3) and twelve months (T4) after first measurement.
  Interventions: Other: Questionnaire administration
- Control group 1 (No Intervention): Pre-test measures are assessed. Enhanced usual care. Follow-up measures are directly after first consultation (T2) and at three (T3) and twelve months (T4) after first measurement.
- Control group 2 (No Intervention): No pre-test measures are assessed. Enhanced usual care. Follow-up measures are directly after first consultation (T2) and at three (T3) and twelve months (T4) after first measurement.

INTERVENTIONS:
Other: Questionnaire administration — The patient receives the SIPP at two different time points during their RT period. The first time point is before the first consultation with the radiotherapist (before starting RT) and the second time point is before the last consultation with the radiotherapist at the end of the RT period. At both time points, the SIPP is handed over to the radiotherapist at the start of the consultation. The radiotherapist screens the scores of the SIPP to get an overview of potential psychosocial problems and patient's needs of psychosocial care.
  Other Names: Psychosocial assessment; Screening
  Arms: Intervention group 1; Intervention group 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness and feasibility of the Screening Inventory of Psychosocial Problems (SIPP) in consultation settings with respect to early recognition and treatment of psychosocial distress, communication between patients and physicians, and psychological distress and quality of life in cancer patients treated with radiotherapy (RT).

DETAILED DESCRIPTION:
Background: The Screening Inventory of Psychosocial Problems (SIPP) is a short, validated self-administered questionnaire to identify psychosocial problems in cancer patients. The one page 24-item questionnaire assesses physical complaints, psychological complaints, and social and sexual problems. There is very little known about the effectiveness of using the SIPP in consultation settings.

Aim: The aim of this study is to test the hypothesis that using the SIPP may prevent underdiagnosis of early symptoms reflecting psychosocial problems, should facilitate communication between physicians and patients about psychosocial distress and may contribute to adequate referral to relevant psychosocial caregivers.

Methods: A Cluster Randomized Controlled Trail (CRCT) is developed using a Solomon four-group design (two intervention and two control groups) to evaluate the effects of using the SIPP. Radiotherapists instead of patients are at random allocated to experimental or control groups. All included patients are randomized into the groups with and without pre-measurement. Psychosocial distress, quality of life, patients' satisfaction about communication with their radiotherapist during first consultation and the number and type of referred patients to psychosocial caregivers are assessed. Self-administered assessments are conducted at four times: pre-test before first consultation (T1), and post-tests directly following the first consultation (T2), three months (T3) and one year after (T4) the first measurement. Medical information are gathered from patients' medical records. Furthermore, a process evaluation is carried out.

Relevance: Using the SIPP may lead to a reduction of psychosocial problems and better quality of life, both on the short and long term. If the SIPP proves to be effective, the results of this project may contribute to motivate health care workers to use the SIPP as a standard method for early detection of psychosocial distress in oncology departments in the Netherlands and abroad.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer
* Lung Cancer
* Prostate cancer
* Bladder Cancer
* Colorectal Cancer
* Cervix Cancer
* Cancer of endometrium
* Cancer of Skin
* Hodgkin Lymphoma
* Non-Hodgkin Lymphoma
* Must receive radiotherapy treatment (RT)
* 18 years of age or older

Exclusion Criteria:

* Metastases
* Less than 10 fractions of radiotherapy treatment (RT)
* Unable to read, and speak Dutch
* Unable to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary effect outcome measurement is the number and type of referred patients with psychosocial problems to psychosocial caregivers and type of referrals with respect to psychosocial problems. | Is measured at three (T3) and twelve (T4) months after first measurement

SECONDARY OUTCOMES:
The secondary outcome measurements are patients' satisfaction with the radiotherapist-patient communication, psychosocial distress and quality of life. | Patients' satisfaction with the radiotherapist-patient communication is measured after first consultation with radiotherapist (T2) and psychosocial distress and quality of life is measured at three (T3) and twelve months (T4) after first measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Lechner, PhD, Principal Investigator — Netherlands Open University, Faculty of Psychology; Gertrudis I Kempen, PhD, Principal Investigator — Maastricht University, Faculty of Health, Medicine, and life Sciences, Department of Health Care and Nursing Science, School for Public Health and Primary Care (CAPHRI)
Locations (1):
- Institute Verbeeten, Tilburg, North Brabant, Netherlands

REFERENCES:
- [Derived] Braeken AP, Kempen GI, Eekers D, van Gils FC, Houben RM, Lechner L. The usefulness and feasibility of a screening instrument to identify psychosocial problems in patients receiving curative radiotherapy: a process evaluation. BMC Cancer. 2011 Nov 8;11:479. doi: 10.1186/1471-2407-11-479. PMID 22067707
- [Derived] Braeken AP, Lechner L, van Gils FC, Houben RM, Eekers D, Ambergen T, Kempen G. The effectiveness of the Screening Inventory of Psychosocial Problems (SIPP) in cancer patients treated with radiotherapy: design of a cluster randomised controlled trial. BMC Cancer. 2009 Jun 9;9:177. doi: 10.1186/1471-2407-9-177. PMID 19508716